# Consent

Official Title of Record: Propylene Glycol-Free Melphalan HCI (EVOMELA®) in Combination with Fludarabine and Total Body Irradiation Based Reduced Intensity Conditioning for Haploidentical Transplantation

NCT03159702

March 28, 2023

**Informed Consent for Research** 

Clinical Interventions template - Version: March 30, 2018

IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

# Medical College of Wisconsin and Froedtert Hospital INTRODUCTION TO THE INFORMED CONSENT

| Name of Subject: |
|------------------|

A Phase II, Open-Label, Study of Propylene Glycol-Free Melphalan for Injection (EVOMELA®) in Combination with Fludarabine and Total Body Irradiation Based Reduced Intensity

Conditioning for Haploidentical Transplantation

Mehdi Hamadani, MD
Froedtert Hospital & the Medical College of Wisconsin
Division of Hematology and Oncology
9200 W. Wisconsin Avenue
Milwaukee WI 53226
414-805-6700

You are invited to take part in this research. You can decide whether to take part in this project or not. You are free to say yes or no. If there is anything that you do not understand, please ask questions.

## **Definitions**

Haplo Identical Hematopoietic Cell Transplantation: A type of allogeneic transplant. It uses healthy, blood-forming cells from a half-matched donor to replace the unhealthy ones. The donor is typically a family member.

Reduced Intensity Conditioning: Reduced intensity conditioning refers to a conditioning regimen that uses less chemotherapy and radiation than the standard myeloablative conditioning.

Immunosuppression Therapy: Treatment that lowers the activity of the body's immune system.

GVHD: Graft versus Host Disease: a complication that can occur after an allogenic bone marrow transplant


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

## **Purpose**

This project is being done to find out more about the safety and tolerability of reduced intensity conditioning (RIC) consisting of Propyhlene Glycol-Free Melphalan for Injection (EVOMELA®) in combination with Fludarabine and Total Body Irradiation (TBI).

## Length

You will be in this research project for about 2.5 years or until progression with two years additional follow-up.

## **Procedures**

## List of visits:

Baseline Visit

- Total Number: 1

Total Time: approximately 3 to 6 hours

Days on which Drugs Are Given

- Total Number: 5

- Total Time: approximately 3 to 5 hours

Irradiation

- Total Number: 1

- Total Time: approximately 2 hours

Transplant Day

- Total Number: 1

- Total Time: approximately 3

hours

 Follow-up Visits Post-transplant Evaluation

- Total Number: 6

- Total Time: approximately 1 to 2

hours

# Procedures that will occur at various visits:

## **Invasive Procedures**

- Transplant, blood draws, total body irradiation.

# **Non-invasive Procedures**

- Physical exam, CT/PET, lung function tests, echocardiogram.

# **Risks**

This is a brief list of the most commonly seen side effects. The *full consent form* after this introduction contains a more complete list of potential research risks.

# Drug risks:

#### **EVOMELA®**

- · Loss of appetite
- Vomiting
- Fatigue
- Constipation
- Diarrhea

#### Fludarabine

- · Low blood counts
- Infection
- Nausea

## Total Body Irradiation (TBI)

- Diarrhea
- Nausea
- Stomach Cramps

# **Bone Marrow Transplant (BMT)**

- Graft rejection
- Slow recovery of blood counts (the red blood cells, white blood cells, and platelets can be slow to recover after transplant)
- Organ Failure including heart, kidney, lung, brain, liver or other body parts

#### Cyclophosphamide

- Sores in mouth or on lips
- Damage to male (testies) and female (ovaries) sex glands
- Infertility

## Mycophenolate Mofetil (MMF)

- Nausea
- Low White Blood Cell count and increased risk of infection
- · Low Platelet count and increased risk of bleeding
- Low red blood cell count and increased need for red cell transfusions

#### **Tacrolimus**

- Kidney problems
- Loss of magnesium, calcium, potassium
- High blood pressure


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

# **Benefits**

We don't know if this project will help you. Your condition may get better but it could stay the same or even get worse.

# **My Other Options**

You do not have to join this project. Your other options may include:

- Joining a different project
- Routine care for this condition
- Getting no treatment for this condition

If you have more questions about this project at any time, you can call Mehdi Hamadani, MD, at 414-805-6700.

If you have questions about your rights as a participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

## **CONSENT TO PARTICIPATE IN RESEARCH**

## A1. INTRODUCTION - WHY ARE WE ASKING YOU TO PARTICIPATE?

You are being invited to participate in this research study because you have a blood cancer and you will be receiving a Haplo Identical Hematopoietic Cell Transplantation (Haplo-HCT).

A total of about 43 people are expected to participate in this research at the Medical College of Wisconsin/Froedtert Hospital/Froedtert Hospital.

The Director of the project is Mehdi Hamadani, MD in the Department of Medicine. A research team works with Dr. Hamadani. You can ask who these people are.

Spectrum Pharmaceuticals, Inc., provides financial support to the Medical College of Wisconsin, including Dr. Hamadani for the work on this study. Dr. Hamadani is the sponsor of the study.

## A2. DO I HAVE TO PARTICIPATE?

You can decide whether to take part in this research or not. You are free to say yes or no. If you say no, your regular medical care will not change. Even if you join this project, you do not have to stay in it. You may stop at any time.

A research project is different from routine medical care in three ways: 1) there are extra risks that we will tell you about in this form; 2) you may have some extra medical tests and visits; 3) the research procedures, tests and visits follow a set plan that must be kept.

# A3. WHY IS THIS PROJECT BEING DONE?

In this study, we want to find out the safety and tolerability of reduced intensity conditioning (RIC) consisting of Propyhlene Glycol-Free Melphalan for Injection (EVOMELA®) in combination with Fludarabine and Total Body Irradiation (TBI) for subjects undergoing Haplo Identical (which involves matching your tissue type with a related or unrelated donor) Hematopoietic Cell Transplantation (Haplo-HCT).

Total Body Irradiation (TBI) is radiation of the entire body as part of the conditioning portion of the study.

Propylene Glycol-Free Melphalan for Injection (EVOMELA®) (study drug) is a combination of melphalan (active drug) and Captisol® (inactive ingredient) that that will be administered by intravenous (IV). This Melphalan formulation does not contain the propylene glycol solvent found in the Melphalan product given as the current standard of care and researchers hope this will lead to improvements for patients. This combination of Melphalan and Captisol® has been approved by the United States Food and Drug Administration (FDA) for treatment in multiple myeloma patients.

For the remainder of this consent, we will refer to the study drug as EVOMELA®.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

## **B1. WHAT WILL HAPPEN IF I PARTICIPATE**

If you choose to take part in this study, you will be asked to sign this consent form. Your study doctor will check your general health to assure that you are eligible to participate in the study. Many of the tests and procedures listed below are part of your regular care. You may have had some of them done already.

# **Screening Period (prior to transplant):**

- Medical history and a review of your current medications
- Physical Examination including your height, weight, and your performance status (your general strength and ability to carry out your daily activities)
- Vital signs including blood pressure, pulse rate, breathing rate and temperature
- Routine blood tests:
  - To check your blood counts (CBC), chemistries, liver function, and kidney function
  - To check for CMV, hepatitis A, hepatitis B, hepatitis C, HIV testing, EBV infection and herpes simplex virus infection
  - o To check your current immune system
  - o To check for pregnancy if you are a woman of childbearing potential
- A MUGA scan or Echocardiogram (ECHO) to test your heart function
- PET/CT
- Lung (pulmonary) function tests

If the screening information shows that you meet the requirements of this research study, then you will be able to start the study. If the screening information shows that you cannot be in the research study, the study doctors will discuss other options with you and/or refer you back to your regular doctor.

# **Conditioning (pre-transplant chemotherapy and radiation):**

You will get drugs and radiation to suppress the immune system and destroy the abnormal marrow, so the donor's healthy cells can grow and produce new blood cells. This is called "conditioning." You will get these drugs through the central venous catheter:

## If you are <60 years old-

- EVOMELA®: (IV) 140mg/m² prior to your bone marrow transplant (BMT) on Day -6
- Fludarabine-: IV 40mg /m² infused over 30 minutes given prior to your BMT on Days -5, -4, -3, -2
- TBI: 200 cGy prior to your BMT on Day -1

For patients who are ≥60 years and/or HCT-CI score of >3 (at the discretion of treating physician will have an option to receive):-

- EVOMELA®: 70 mg/m²/day IV on Day -6
- Fludarabine: IV 40 mg/m²/day infused over 30 minutes given prior to your BMT on Days -5, -4, -3, -2
- TBI: 200 cGy on Days -1


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

# **EFFECTIVE**

3/28/2023

MCW/FH IRB

## **Study Procedures**

# Day -6 through Day -1 (prior to transplant)

- Physical Examination (your general strength and ability to carry out your daily activities)
- Vital signs including blood pressure, pulse rate, breathing rate and temperature
- Blood tests:
  - To check your blood counts (CBC), chemistries, liver function, and kidney function

# Day 0 (transplant)

You will receive the donor's bone marrow stem cells.

The following will also be completed:

- Physical Examination (your general strength and ability to carry out your daily activities)
- Vital signs including blood pressure, pulse rate, breathing rate and temperature
- Blood tests:
  - To check your blood counts, chemistries, liver function, and kidney function
  - o To check for CMV EBV infection and herpes simplex virus infection

# **Immunosuppression Therapy**

As part of the standard transplant procedure, you will be given drugs to reduce the risk of graft versus host disease (GVHD), a complication that occurs when the donor blood cells recognize the body as foreign and attack it. These drugs are usually started around the time you receive the donor cells and can continue many months after the transplant. The drugs do not completely prevent GVHD and more drugs might be needed if you do develop GVHD.

Below is a list of the drugs commonly used that you will receive to prevent GVHD:

- Tacrolimus
- Mycophenolate Mofetil (MMF)
- Cyclophosphamide

## **Post-Transplant Care**

As part of the standard transplant procedure you will stay in the hospital until your white blood count has returned to acceptable levels and you are able to take your medications by mouth. While in the hospital you will have daily blood tests that require 2–3 tablespoons of blood. You may also have other tests or procedures that the study doctor (your transplant doctor) and team think are necessary to monitor your health. You will be watched for any side effects from the drugs or the transplant itself. You will be given drugs and/or treatment to lessen any side effects that may occur.

## **Post-Transplant Evaluations**

As part of the standard transplant procedure, you will have blood drawn at specific time points. Bone marrow examinations will be performed as determined by your doctor to meet standard of care needs. These tests are to evaluate how your new blood cells are developing and how your immune system is recovering after the transplant. We will also be testing what fraction of the blood is made up of donor or your cells after the transplant.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

You will be discharged from the inpatient bone marrow transplant unit when you are ready to be cared for as an outpatient. After discharge you will be seen by the transplant doctor and team in the bone marrow transplant clinic at least weekly for follow-up. Usually the frequency of office visits will decrease three months after the transplant, but this will depend on how well you are doing.

We would like to continue to follow you for a total of two years after your transplant for disease status and survival. We will talk to you about any side affects you may have experienced during this study at your normal clinic visits or hospital stays. Your follow-up visits during the first two years is no more frequent than standard for most patients at our center.

Infectious Disease Testing

As part of the procedure for donating a unit of blood, your blood will be tested for diseases that can be passed on to other people by transfusion, including AIDS (the disease caused by the HIV virus), hepatitis B, hepatitis C and others. If certain tests are positive, wemay inform you, and inform certain government health agencies as required by law. Results of your blood test will be released only to authorized persons as governed by Wisconsin law. A list of persons to be notified and reasons that will cause release of your blood test is available upon request. Results of the blood test will be released to Versiti, Inc. physicians and their assistants, and the study team members and staff.

## **B2. HOW LONG WILL I BE IN THE PROJECT?**

You will be in this research study for about 2.5 years or until progression, with two years additional follow-up.

#### **B3. CAN I STOP BEING IN THE PROJECT?**

You are free to withdraw from the project at any time. If you leave, your regular medical care will not change. If you are thinking about leaving, please tell the research doctor.

- ⇒ The research doctor can tell you about the effects of stopping, and you and the research doctor can talk about what follow-up care would help you the most.
- ⇒ You might be asked to come back for one more visit to check your health.

The research doctor may take you out of this project at any time. This would happen if:

- They think it is in your best interest.
- You do not follow the project rules.
- The whole project is stopped.

If this happens, the research doctor will tell you.

## C1. WHAT HEALTH RISKS OR PROBLEMS CAN I EXPECT FROM THE PROJECT?

There are risks to taking part in any research project. There is a risk that you may get a drug/drug combination that does not help your condition or may make it worse. There also may be problems (side effects) we do not know about yet, from the drugs themselves, or how it combines with other drugs you are taking. If we learn about new important side effects, we will tell you.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

We watch everyone in the project for problems (side effects). You need to tell the research doctor or a member of the research team immediately if you experience any problems, side effects, or changes in your health. If you have problems, call Dr. Hamadani immediately at 414-805-6700. In an emergency, call 911.

# C2. RISKS OF RESEARCH TREATMENT

The research/intervention itself may cause problems (side effects). Side effects may be mild or very serious. Some can last a long time or never go away. Many go away soon after you stop taking the drugs. Drugs can affect individuals in different ways. Complications of some of the side effects below may lead to life-threatening events and possibly death.

The risks of the drugs you will get as part of the treatment are listed below.

# **EVOMELA®**

# Likely (May happen in more than 20% of patients)

- Loss of appetite
- Vomiting
- Fatigue
- Constipation
- Diarrhea
- Nausea (feeling sick to your stomach)
- Temporary hair loss
- Sensitive skin
- Infection
- Low number of white blood cells
- Low number of platelets in the blood with increased risk of bleeding
- Anemia (low number of red blood cells)
- Mouth sores
- Sore throat (red with swelling)

## Less Likely (May happen in less than 20% of patients)

- Changes in heart beat
- Dizzy
- Feeling faint
- Shortness of breath
- Hepatitis (swelling of the liver)
- Kidney failure
- Weight loss
- Feeling weak


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

# Rare but Serious (May happen in less than 2% of patients)

- Allergic reaction
- Lung infection
- Scarring of lung tissue
- Seizure
- Vasculitis (inflammation of blood vessels)
- Low blood pressure
- Sweating too much
- Sterility (unable to have children
- Liver damage
- New cancer of bone marrow cells

# **Fludarabine**

# Likely (May happen in more than 20% of patients)

- Low blood counts
- Infection
- Nausea
- Vomiting
- Diarrhea

# Less Likely (May happen in less than 20% of patients)

- Fever
- Numbness in the extremities
- Sleepiness
- Visual Changes
- Weakness
- Fatigue

# Rare but Serious (May happen in less than 2% of patients)

- Coma
- Cough
- Skin rash
- Inflammation of the lung
- Interstitial Pneumonia (type of lung disease)
- Neurotoxicity, including blindness, coma, weakness, agitation, visual disturbances, and death
- Secondary Cancers

# **Total Body Irradiation (TBI)**

## Likely (May happen in more than 20% of patients)

Diarrhea


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

- Nausea
- Stomach Cramps
- Vomiting
- Painful swelling of the parotid gland (salivary glands under the ears) for a few days
- Short-term hair loss
- Anemia
- Infection
- Bleeding
- Cataracts
- Sterility (inability to have children)
- Growth failure
- Endocrinopathies (such as thyroid disease or diabetes)
- Mouth sores

## Less Likely (May happen in less than 20% of patients)

- Lung inflammation
- Pneumonia
- Redness of the skin
- Liver problems

# Rare but Serious (May happen in less than 2% of patients)

- Risk of developing other cancers in the future as a consequence of having received the total body irradiation
- Difficulty swallowing
- Back problems
- Kidney problems

## **Bone Marrow Transplant (BMT)**

- Graft rejection
- Slow recovery of blood counts (the red blood cells, white blood cells, and platelets can be slow to recover after transplant)
- Organ Failure including heart, kidney, lung, brain, liver or other body parts
- Acute GVHD
  - Skin rash
  - Nausea
  - Vomiting
  - o Diarrhea
  - Abdominal (stomach area) pain
  - o Problems with your liver (your doctor will run tests for this
  - o Infection
- Chronic GVHD
  - Skin rash


Version: MCW v43-28-2023

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

3/28/2023

**EFFECTIVE** 

MCW/FH IRB

- Hair loss
- Thickened skin
- Joint stiffness (knees, elbows, fingers)
- o Dry eyes
- Dry mouth
- Liver disease (your doctor will run tests for this)
- Weight loss
- Diarrhea
- Infection

# Cyclophosphamide

# Likely (May happen in more than 20% of patients)

- Sores in mouth or on lips
- Damage to male (testis) and female (ovaries) sex glands
- Infertility
- Irregular or no menstrual cycles
- Diarrhea
- Fluid retention
- Alopecia (hair loss)
- Nausea
- Vomiting
- Headache
- Loss of appetite
- Suppression of immune system
- Decreased platelet count and increased risk of bleeding

## Less Likely (May happen in less than 20% of patients)

- Bleeding in bladder
- Anemia (low red blood cell count)
- Damage to the fetus if you become pregnant while taking drug
- Stomach pain
- Skin rash

# Rare but Serious (May happen in less than 2% of patients)

- Allergic reaction
- Lung fibrosis (scarring of lung tissue with cough and shortness of breath)

## Mycophenolate Mofetil (MMF)

## Likely (May happen in more than 20% of patients)

- Nausea
- Low White Blood Cell count and increased risk of infection


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

- Low Platelet count and increased risk of bleeding
- Low red blood cell count and increased need for red cell transfusion

# Less Likely (May happen in less than 20% of patients)

- Vomiting
- Diarrhea
- Rash
- Sleeplessness
- Leg Cramps
- Bone pain
- Changes in blood chemistry
- Headaches

# Rare but Serious (May happen in less than 2% of patients)

- Infection of the brain
- Risk to a baby in pregnancy
- Secondary cancers, such as lymphoma or lymphoproliferative disease
- Hypertension

# **Tacrolimus**

# Likely (May happen in more than 20% of patients)

- Kidney problems
- Loss of magnesium, calcium, potassium
- High blood pressure
- Tremors
- Increases in cholesterol and triglyceride
- Decreased platelet count with increased risk of bleeding
- Infections

# **Less Likely (May happen in less than 20% of patients)**

- Nausea
- Vomiting
- Liver problems
- Changes in how clearly one can think
- Insomnia
- Unwanted hair growth
- Confusion

# Rare but Serious (May happen in less than 2% of patients)

- Seizures
- Changes in vision


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

Dizziness

Red blood cell destruction

MCW/FH IRB

**EFFECTIVE** 

3/28/2023

It is very important that you do not eat grapefruit or drink grapefruit juice while taking Tacrolimus. Grapefruit has an ingredient called bergamottin, which can affect some of the treatment drugs used in this study. Common soft drinks that have bergamottin are Fresca, Squirt, and Sunny Delight.

## C3. OTHER RISKS OF THIS RESEARCH PROJECT

Other procedures and medications that are part of the research also involve some risks:

# **Blood Drawing**

The risks of drawing blood from a vein include discomfort at the site of puncture (where the needle is placed in the vein); possible bruising and swelling around the puncture site; rarely, an infection; and uncommonly, faintness from the procedure.

# **Bone Marrow Aspiration and Biopsy**

A bone marrow aspiration is a procedure in which an area of the hip (buttock area) is numbed with local anesthetic, and a small sample of bone marrow is withdrawn. A bone marrow biopsy is similar to a bone marrow aspiration, except a sample of bone is removed through the needle. When the local anesthesia is given, you may initially feel a burning sensation in your skin and bone surface for several seconds. During the actual procedure itself, you may temporarily feel pressure and/or pain of varying degrees. If necessary, you may ask your physician for additional local anesthesia or a medication to ease your stress. You also may experience bleeding, and/or bruising after the procedure is completed and you may experience soreness in the area for a few days afterwards. Rarely an infection can develop.

## CT/PET Scan

A CT scan is a test that uses a small amount of radiation (x-ray) to make pictures of the inside of your body. For this test, the study doctor or research staff may give you a contrast dye, either by mouth or with a needle. You may feel a sharp sting when the needle is placed in your vein followed by a feeling of warmth throughout the body.

There is a slight risk of developing an allergic reaction to the contrast material. Be sure to tell your study doctor if you have allergies of any kind, such as hay fever, iodine allergy, eczema, hives, or food allergies. There is always a slight risk from being exposed to any radiation, including the low levels of x-rays used for a CT scan. However, the risk from the x-rays is usually very low compared with the potential usefulness of the test to manage your treatment. Confinement and claustrophobia may be experienced during the scan.

A PET scan uses a small amount of radioactive material (tracer). The tracer is given through a vein (IV). The needle is most often inserted on the inside of your elbow. The tracer travels through your blood and collects in organs and tissues. This helps the radiologist see certain areas more clearly. You may feel a sharp sting when the needle with the tracer is placed into your vein. Rarely, people may have an allergic reaction to the tracer material. Some people have pain, redness, or swelling at the injection site.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

# **Echocardiogram (ECHO)**

The ECHO involves placing a gel on the skin of the chest and rubbing the ultrasound wand over your heart to see the blood pumping out of your heart. There are no known complications from the ECHO procedure.

## **MUGA**

The MUGA involves injecting a small amount of imaging agent (radioactive tracer) into a vein in your arm and then scanning. The tracer and the scan let the doctor see how well the chambers of your heart pump blood. The level of radiation is very low. You may have an allergic reaction to the tracer.

## **C4. REPRODUCTIVE RISKS**

# Risks to women who could become pregnant

The drugs in this project might affect a baby, before or after the baby is born. We do not know if the drugs cause harm to a baby, so we do not want anyone who might be pregnant to enter the project. You should not become pregnant or nurse a baby while in this project. You must tell the research doctor right away if you think you are pregnant. You will be asked to have a pregnancy test to be sure you are not pregnant at the start of the project.

# Risks of fathering a child

You should not father a baby while taking part in this project because it is unknown if the drugs could affect a baby. If your partner is able to become pregnant, one or both of you must use some form of effective birth control. You must tell the research doctor right away if you think your partner is pregnant.

# Birth control methods for all subjects

Check with the research doctor about the birth control methods needed for this project and how long to use them. Some methods might not be good enough for this project. If you are having sex that could lead to pregnancy, you should use birth control while you are in this project. This may include:

- Not having vaginal sex (abstinence)
- Taking birth control pills orally
- Having birth control shots or patches such as Depo-Provera
- Surgical sterilization (hysterectomy or tubal ligation)
- Use of an intrauterine device (IUD)
- Use of diaphragm with contraceptive jelly
- Use of condoms with contraceptive foam
- Use of diaphragm with condoms ("double barrier")
- Limiting sexual activity to a male partner who has had a vasectomy

You should use two effective methods of birth control at the same time from the time you sign consent through 90 days after the last dose of the study drug and must also adhere to the guidelines of any treatment-specific pregnancy prevention program.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

## C5. ARE THERE ANY BENEFITS TO TAKING PART IN THE PROJECT?

We don't know if this study will help you. Your condition may get better but it could stay the same or even get worse. We hope the information from this study will help us develop better treatments for blood cancers.

## D1. ARE THERE ANY COSTS TO BEING IN THE PROJECT?

Most of the medical care that you will receive in this study is considered routine care for your condition and would be recommended whether you join the study or not. Costs for routine care will be billed to you or your insurance carrier.

Activities / costs that are part of the study will not be billed to you or your insurance company. This is the study drug, EVOMELA®. Some insurers will not pay for drugs, tests or hospitalization that are part of research studies, so check with your insurer before you join this study. If you have questions regarding study costs, please contact Dr. Hamadani.

If you participate in this research, the costs of any necessary emergency medical treatment in the event of a research-related injury will be billed to you or your health insurance.

## D2. WILL I BE PAID FOR PARTICIPATING IN THE PROJECT?

There is no payment for being in this study.

## D3. WHAT OTHER HEALTHCARE CHOICES DO I HAVE?

You do not have to join this project. You are free to say yes or no. If you do not join this project, your research doctor can discuss other healthcare choices with you. Your other choices may include:

- You may receive melphalan in its standard form
- Joining a different research study
- Getting treatment or care for your cancer without being in a study.
- Getting no treatment
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

The research doctor can explain both the possible benefits and the risks of other options that are available to you.

## D4. WILL I BE GIVEN NEW INFORMATION ABOUT THE PROJECT?

If we learn any important new information about the drug that might change your mind about being in the project, we will tell you about it right away. You can then decide if you want to stay in the project.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

When research data is collected and analyzed, there is the chance of finding something clinically relevant. There may be benefits to learning such results (such as early detection and treatment of a medical condition), but there are risks as well (such as feeling worried about a finding for which no treatment is required or appropriate).

The results from the data we collect in this research study are not the same quality as what you would receive as part of your health care, so you will not be informed of any clinically relevant research findings. The results of your research data will not be placed in your medical record.

## D5. WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THE PROJECT?

Emergency medical treatment for injuries directly related to your participation in this research project will be provided to you. You or your health insurance will be billed for the costs of this emergency treatment. MCW will decide on a case by case basis if they will reimburse you or your insurer for emergency treatment costs. If your research-related injury requires medical care beyond this emergency treatment, you or your insurer will be responsible for the costs of this follow-up care.

At this time, there is no plan for any additional financial payments.

If you believe that you have been injured because of your participation in this project, contact the research doctors right away. Contact information: Dr. Hamadani at 414-805-6700.

Nothing in this consent form affects any legal rights you may have nor does it release the investigator, the sponsor, the institution, or its agents from liability for negligence.

## D6. WHO CAN ANSWER MY QUESTIONS ABOUT THE PROJECT?

- If you have more questions about this project at any time, you can call Dr. Hamadani at 414-805-6700.
- If you have questions about your rights as a research participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.

# E. PERMISSION TO COLLECT, USE AND SHARE HEALTH INFORMATION

# E1. What health information will be collected and used for this project?

To be in this research project, the research team needs your permission to access, collect and use some of your health information. If you say no, you cannot be in the project. This information may come from questions we ask, forms we ask you to fill out, or your medical record, as described below. We will only collect and use information needed for the project.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

The protected health information (PHI) originates from services you will or have received at one or more of the following locations: the Medical College of Wisconsin (MCW); BloodCenter of Wisconsin (BCW); Children's Hospital of Wisconsin (CHW); any Froedtert Health Affiliate-Froedtert Memorial Lutheran Hospital (FMLH), Inc.; Community Memorial Hospital (CMH) Menomonee Falls, Inc.; St. Joseph's Community Hospital (SJH) West Bend, Inc.; Froedtert & The Medical College of Wisconsin Community Physicians Clinics, Inc. (FMCWCP); the West Bend Surgery Center, LLC; and the Froedtert Surgery Center, LLC.

# The health information to be collected and used for this project is:

- Hospital/Medical Records
- Physician/Clinical Records
- Lab and/or Pathology Reports
- Radiology Reports
- Biological Samples

# E2. Who will see the health information collected for this project?

The only MCW/Froedtert Hospital employees allowed to handle your health information are those on the research team, those on the Institutional Review Board (IRB) and those who check on the research activities to make sure the hospital's rules are followed.

If the costs of any necessary emergency medical treatment in the event of a research-related injury are billed to your health insurance, your health information may need to be disclosed to the insurer for billing purposes.

The research team may share your information with people who don't work at MCW/Froedtert Hospital because they planned, pay for, or work with us on this project. The federal Privacy Rule may no longer protect your health information once it leaves MCW/Froedtert Hospital. For this project, we plan to share information with those doctors, researchers or government representatives working with us on this project at the institutions or companies listed here:

- Spectrum Pharmaceuticals, Inc.
- U.S. Food and Drug Administration (FDA), Rockville, MD
- Federal agencies such as the Department of Health and Human Services (the DHHS), the National Cancer Institutes / National Institutes of Health (the NCI/NIH) and the Office for Human Research Protections (the OHRP)
- Any independent ethics committee, which approved this study
- Those required by law
- Florence Healthcare Inc.

Because this project involves the use of drugs and/or devices, the FDA also has the right to inspect all project records.


Medical College of Wisconsin & Froedtert Hospital **Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 – 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

We may record your research information, including results of tests and procedures done for research, in your Froedtert Hospital and/or Medical College of Wisconsin medical record. As a result, this research information may be seen by people allowed to see your medical records for healthcare operations or treatment, by those you allow to see your medical records by giving written permission, and by others when required by law.

We will not use your personal health information for a different project without your permission or the permission of a hospital research review board (IRB). Once all personal identification is removed from your health information and/or biospecimens, the information and/or biospecimens may be used for future research or distributed to another investigator for future research without additional informed consent from you or your legally authorized representative. The information might also be used or released for other purposes without asking you. Results of the project may be presented in public talks or written articles, but no information will be presented that identifies you.

# E3. What are the risks of sharing this health information?

One risk of taking part in a research project is that more people will handle your personal health information collected for this project. The research team will make every effort to protect the information and keep it confidential, but it is possible that an unauthorized person might see it. Depending on the kind of information being collected, it might be used in a way that could embarrass you or affect your ability to get insurance. If you have questions, you can talk to the research doctor about whether this could apply to you.

# E4. How long will you keep the health information for this project?

If you sign this form, we plan to keep your information without any end-date in case we need to check it again for this project.

## E5. Can I cancel my permission to share this health information?

If you change your mind later and do not want us to collect or share your health information, you need to send a letter to Dr. Hamadani at:

Mehdi Hamadani, MD Froedtert & Medical College of Wisconsin Division of Hematology and Oncology 9200 W. Wisconsin Avenue Milwaukee, WI 53226

The letter must say that you have changed your mind and do not want the researcher to collect and share your health information. At that time, we may decide that you cannot continue to be part of the project. We may still use the information we have already collected.

## E6. Access to records

You may not be able to see, or copy, your project-related health information until after the project has been completed; otherwise, it could affect the study.


Medical College of Wisconsin & Froedtert Hospital **Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

# F1. FOR MORE INFORMATION ABOUT THE PROJECT

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can look up this project by referring to the ClinicalTrials.gov number (NCT03159702) or by asking the research team for a printed copy.


**Informed Consent for Research** 


IRB Protocol Number: 29507

IRB Approval Period: 3/28/2023 - 3/27/2024

**EFFECTIVE** 

3/28/2023

MCW/FH IRB

# **CONSENT TO PARTICIPATE**

# By signing my name below, I confirm the following:

- I have read (or had read to me) this entire consent document. All of my questions have been answered to my satisfaction.
- The project's purpose, procedures, risks and possible benefits have been explained to me.
- I agree to let the research team use and share the health information and other information gathered for this project.
- I voluntarily agree to participate in this research project. I agree to follow the procedures as directed. I have been told that I can stop at any time.

**IMPORTANT:** You will receive a signed and dated copy of this consent form. Please keep it where you can find it easily. It will help you remember what we discussed today.

| Subject's Name please print | Subject's Signature | Date |
|---|---|---|
| Name of Witness please print | Signature of Witness | Date |
| Rationale for Use of Witness | | |
| ☐ Subject has limited/no literacy | ☐ Sponsor requirement | |
| Subject has limited English | Other | _ |
| proficiency | | |
| ☐ Subject has limited/no vision | | |
| * Name of person discussing/<br>obtaining consent please print | Signature of person discussing/obtaining consent | Date |


<sup>\*</sup> A member of the research team trained and authorized by the Principal Investigator to act on her/his behalf in obtaining informed consent according to the protocol. The Principal Investigator is responsible and accountable for the research project.